CLINICAL TRIAL: NCT04932720
Title: Efficacy of Child Yoga Programme on Quality of Life of Pediatric Oncology Patients.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, N.Ecem Oksal Gunes, Phd, Principal investigator, Cukurova University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 11814
Record Dates: First submitted 2021-06-08; First posted 2021-06-21 (Actual); Last update posted 2021-08-13 (Actual); Status verified 2021-06

CONDITIONS: Pediatric Cancer
Keywords: Child Health and Diseases Nursing; cortisol; quality of life; stress; yoga
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: Children who were treated at Mersin University Medical Faculty Hospital were determined by the "simple random selection" method and formed the experimental and control groups.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): Experimental group consisted of children aged 8-18 years, who did not have a different disease accompanying the oncological disease.
  Interventions: Behavioral: chıld yoga programme
- control group (No Intervention): Also the control group consisted of children aged 8-18 years, who did not have a different disease accompanying the oncological disease.

INTERVENTIONS:
Behavioral: chıld yoga programme — Yoga sessions were in the form of 6 sessions and were held as 2 sessions per week. The program was given by an expert yoga instructor who has an international "Yoga Alliance" approved child and adolescent yoga certificate.Consisting of the components of Hatha Yoga (HY), one of the yoga types known and widely practiced all over the world; Sessions consisting of asanas (yoga postures), pranayamas (breathing techniques), relaxation, relaxation exercises and meditation were prepared. Sessions are 45 minutes; For those who are new to yoga for the first 15 minutes; mental and physical preparation; asanas, pranayamas were taught, drama followed by breathing exercises and asanas in the next 30 minutes, relaxation techniques (imaginary journey) and meditation in the last 15 minutes.
  Arms: experimental group

SUMMARY:
Pediatric oncology patients experience physical and psycho-social symptoms that negatively affect their quality of life during treatment. "Yoga" practices, known as a unique physical activity that combines mind-body awareness and breathing exercises to improve the quality of life of pediatric oncology patients, have recently become popular.

The study was conducted experimentally in the form of pre-test and post-test with 30 controls, 30 experimental group children who were treated in the Pediatric Oncology / Hematology service of a university hospital and their parents, in order to investigate the effect of children's yoga program on the quality of life of pediatric oncology patients. Ethics committee, institutional and parental consent was obtained. Data were collected using a questionnaire form and the Pediatric Quality of Life Inventory "PedsQL (4.0)". Participants filled out the Pediatric Quality of Life Inventory "PedsQL (4.0)" Child and Parent Form before the 3-week (6 sessions) yoga program and salivary cortisol samples were taken from the children. These procedures were repeated after the yoga program. Anova test and "Paired sample t" test were used among statistical analysis methods. Statistical significance was accepted as p <0.05.

DETAILED DESCRIPTION:
A questionnaire form was used to learn the socio-demographic characteristics of the children participating in the study and their families. The survey questions are: (age of parents, employment status, child's age, gender, maternal/paternal age, income status, diagnosis of the child, hospitalization the reason (chemotherapy, new diagnosis, relapsed? hospitalized for side effects of the disease? how much whether he was diagnosed a long time ago, how long he has been in the hospital, whether he went to school, whether he had previous yoga experience, whether he had knowledge about children's yoga before.

In order to demonstrate the effectiveness of the child yoga program, the study was conducted with pre-test and post-test. Before the first yoga session, the experimental and control group caregiver parents and children was completed the quality of life inventory.

The children's yoga program lasted for 3 weeks, 2 sessions per week. At the end of the 6th session, parents and the child's quality of life inventory was repeated.

In order to evaluate the effect of yoga on stress of children, cortisol from saliva samples were taken both groups before the program starts.The measurement was performed for both groups after a 3-week (6 sessions) yoga program.

The hypotheses in the study can be summarized as follows:

H1: Physical activity pre-test and post-test scores of the control and experimental groups There is a significant difference between the groups in favor of the experimental group.

H2: Emotional functionality pre-test and post-test scores of the control and experimental groups there is a significant difference between the groups in favor of the experimental group.

H3: Social functionality pre-test and post-test scores of the control and experimental groups there is a significant difference between the groups in favor of the experimental group.

H4: School functionality pre-test and post-test scores of the control and experimental groups there is a significant difference between the groups favor of the experimental group.

H5: Cortisol levels, pre-test and post-test scores of the control and experimental groups there is a significant difference between the groups in favor of the experimental group.

SPSS 22.0 Statistical Package for the Social Sciences program used for data analysis.descriptive, parametric and non-parametric statistical analyzes, mean, standard deviation, median, frequency, percentile, minimum, maximum values calculated. The effectiveness of the yoga program was measured using the anova (mixed anova) test and the "Paired sample t" test. p<0.05 value was accepted as the statistical significance limit.

Chıld Yoga Programme:

In our study, Hatha Yoga, one of the known and widely practiced yoga types all over the world. (HY) consisting of components; asanas (yoga poses), pranayamas (breathing techniques), relaxation, relaxation exercises and meditation sessions were prepared. Sessions are 45 minutes; For those who are new to yoga for the first 15 minutes; mental and physical preparation; asanas, pranayamas taught, drama followed by breathing exercises and asanas in the next 30 minutes, relaxation in the last 15 minutes techniques (imaginary journey) and meditation.

ELIGIBILITY:
Inclusion Criteria:

* Of the participating children, those who did not have any other accompanying disease and did not have developmental disorders were included in the study.

Exclusion Criteria:

* Children who were not approved by the Pediatric Oncology unit responsible doctor for inclusion in the yoga program constituted the limitation of the study.

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2020-01-19 (Actual); Primary Completion 2021-05-19 (Actual); Study Completion 2021-05-19 (Actual)

PRIMARY OUTCOMES:
Quality of Life Inventory (PedsQL 4.0) of 8-12 and 13-18 age were used to evaluate the impact of the child yoga program on quality of life of pediatric oncology patients. | 3 weeks
  A questionnaire form was used to learn the socio-demographic characteristics of the children and their families. Quality of Life Inventory (PedsQL 4.0) of 8-12 and 13-18 age child and parent form were used to evaluate the impact of the child yoga program on quality of life of pediatric oncology patients.It is a versatile inventory of 23 items covering school functions (5 Items), social functions (5 Items), emotional functions (5 Items), physical functions (8 Items). Saliva samples were taken from the experimental and control groups to measure the stress levels of the children with the cortisol kit.

CONTACTS AND LOCATIONS:
Overall Officials: Şenay Çetinkaya, Study Director — Cukurova University
Locations (1):
- Çukurova University, Adana, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No